CLINICAL TRIAL: NCT02279381
Title: A Randomized Controlled Trial to Evaluate the Acceptability, Feasibility and Efficacy of the Use of a Neonatal Package to Reduce Neonatal Infection in a Rural District of Pakistan
Brief Title: Neonatal Package Study in Rural District of Pakistan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: University of Sydney (Other); The International Federation of Red Cross and Red Crescent Societies (Other)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3106-Ped-ERC-14
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Neonatal Infections
Keywords: Chlorhexidine; Kangaroo mother care; RCT
MeSH Terms: interventions — Chlorhexidine; Anti-Infective Agents, Local; Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention group A (Experimental): 1. Essential Neonatal Care
  2. Kangaroo mother Care
  3. Application of 4% Chlorhexidine
  4. Education and counseling for mothers and care providers
  Interventions: Drug: Chlorhexidine; Other: Kangaroo Mother Care; Other: Essential Neonatal Care
- Intervention group B (Experimental): 1. Essential Neonatal Care
  2. Application of 4% Chlorhexidine
  3. Education and counseling for mothers and care providers
  Interventions: Drug: Chlorhexidine; Other: Essential Neonatal Care
- Control group (Active Comparator): 1. Essential Neonatal Care
  2. Education and counseling for mothers and care providers
  Interventions: Other: Essential Neonatal Care

INTERVENTIONS:
Drug: Chlorhexidine — 4% chlorhexidine will be applied to the umbilical stump from day 1 to day 10
  Other Names: Antiseptic
  Arms: Intervention group A; Intervention group B
Other: Kangaroo Mother Care — Skin to Skin Care which is Kangaroo mother care will be carried out by mother from Day 1 till the study completion
  Arms: Intervention group A
Other: Essential Neonatal Care — Essential Neonatal Care ensures delayed bathing, use of colostrum, exclusive breast feeding, skin to skin care for hypothermia, dry cord care, eye care and immunization for the newborn

SUMMARY:
Neonatal mortality has been a notable health issue in Pakistan. Considering the importance of the issue and well recognized interventions the investigators are proposing a randomized controlled trial in a rural district of Pakistan which will evaluate the effectiveness of a neonatal package comprised of the standard neonatal care, Kangaroo Mother Care (KMC) and application of chlorhexidine compared with standard neonatal care coupled with application of chlorhexidine and essential neonatal care alone. The investigators anticipate that this study will provide an evidence base way forward benefiting the children of Pakistan.

DETAILED DESCRIPTION:
The global neonatal mortality burden is one of the imminent factors which derail the achievement of the MDG 4 in many developing countries including Pakistan. Four million infants infants die in their first 28 days of their lives which account for about 40% of the total under-five mortality. The burden of neonatal mortality in Pakistan is alarming as the current neonatal mortality rate (NMR) is 55 per 1000 live births, third worst in the world. The major causes of these deaths are infections, preterm births and birth asphyxia which are avoidable. Despite many initiatives the NMR remains unchanged since last decade in Pakistan.

Literature shows that low cost facility and community based interventions can reduce NMR significantly. Early neonatal care, application of chlorhexidine for cord care and Kangaroo Mother Care (KMC) have been recognized as effective intervention in reduction of neonatal morbidity and subsequently neonatal mortality in many developing countries. However these interventions have never been tested as a package and data about their combined effect is scarce both in Pakistan and developing countries.

Considering the importance of the issue and well recognized interventions we are proposing a randomized controlled trial in a rural district of Pakistan which will evaluate the effectiveness of a neonatal package comprised of the standard neonatal care, KMC and application of chlorhexidine compared with standard neonatal care coupled with application of chlorhexidine and standard neonatal care alone. We anticipate that this study will provide an evidence base way forward benefiting the children of Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* All healthy newborns born in the study settings will be systematically enrolled in the trial after prior consent.

Exclusion Criteria:

* Infants with congenital/birth defects,
* any localized infection on the peri umbilical region at the time of birth or application of
* any other material such as dung etc before enrollment on the cord.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1450 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Reduction in the Incidence of Neonatal infections in the first 28 days of life (Clinical presence of danger signs as per the IMNCI guidelines.) | 28 days post recruitment
  Clinical presence of danger signs as per the IMNCI guidelines.

SECONDARY OUTCOMES:
Reduction in the Incidence of omphalitis (Redness and Swelling of umbilical stump/cord (Inflammation)) | 28 days post recruitment
  Redness and Swelling of umbilical stump/cord (Inflammation):
Failure to thrive (Weight, length and OFC appropriate for age as per WHO guidelines) | 28 days post recruitment
  Weight, length and OFC appropriate for age as per WHO guidelines
Utilization of KMC Compliance, Frequency and duration | 28 days post recruitment
  Compliance, Frequency and duration - hours/day

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Atif Habib, MPH, Study Director — Aga Khan University
Locations (1):
- Taluka Hospital KN Shah, Dadu, Sindh, Pakistan